CLINICAL TRIAL: NCT04433754
Title: Pancreatic Injury in Patients With COVID-19 Disease
Brief Title: The Development of Pancreatic Injury in the Course of Severe Acute Respiratory Syndrome Coronavirus 2 Infection
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Cevdet Duran, Professor, M.D., Uşak University
Other Study IDs: UsakU-Cevdet2
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with pancreatic injury: patients with higher amylase and lipase levels (higher than the laboratory upper limits) in the course of SARS-CoV-2 infection
  Interventions: Other: biochemical analysis
- patients without pancreatic injury: patients with normal amylase and lipase levels in the course of SARS-CoV-2 infection
  Interventions: Other: biochemical analysis

INTERVENTIONS:
Other: biochemical analysis — cRP, d-dimer levels and lymphocyte counts will be compared

SUMMARY:
Although COVID-19 disease due to Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) affects the respiratory tract, heart and coagulation system, symptoms of gastrointestinal system involvement such as abdominal pain, nausea, vomiting and diarrhea are also common.

In this study, it was aimed retrospective analysis of clinical and laboratory data of patients who developed pancreatic injury in the course of COVID 19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with amylase and lipase levels measured during covid-19 disease with or without pneumonia

Exclusion Criteria:

* Patients with pregnancy
* Patients whose amylase and lipase levels were not measured during covid 19 disease
* Patients with known solid organ malignacy
* Patients with known hematologic malignacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who develop amylase and lipase elevation during the course of COVID 19 will be considered in the pancreatic injury group. Those who do not develop will be counted as the control group.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
to compare presence of fever in patients with and without pancreatic injury | 3 month
  To evaluate the frequency of presence of fever in patients with and without pancreatic injury
to compare presence of dyspnea in patients with and without pancreatic injury | 3 month
  To evaluate the frequency of presence of dyspnea in patients with and without pancreatic injury
To compare cRP levels in patients with and without pancreatic injury | 3 month
  CRP levels will be compared in patients with and without pancreatic injury
To compare d-dimer levels in patients with and without pancreatic injury | 3 month
  D-Dimer levels will be compared in patients with and without pancreatic injury

CONTACTS AND LOCATIONS:
Locations (1):
- Usak University Training and Research Hospital, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No